CLINICAL TRIAL: NCT05092659
Title: Patient Experience in Bariatric Surgery: Definition of New Indicators
Acronym: CALEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CALEX; 2021-A02161-40 (Other: ID-RCB)
Record Dates: First submitted 2021-09-22; First posted 2021-10-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient interviews (Other): Patient enrolled in a bariatric surgical pathway scheduled for visceral surgery.
  Interventions: Behavioral: Patient interview

INTERVENTIONS:
Behavioral: Patient interview — Each patient included will be interviewed 3 times : before surgery, 3 and 6 months after surgery

SUMMARY:
Given the growing importance of placing the patient at the heart of care evaluation, the use of patient questionnaires such as Patient Reported Experience Measures (PREMS) or Patient-Reported Outcome Measures (PROMS) has become widespread in recent years. PROMS assess the outcomes of care, whereas PREMS assess the patient's experience of care. However, these tools only imperfectly reflect the patient's experience and only answer specific questions: satisfaction, pain management, waiting times, etc.

Patients undergoing bariatric surgery will undergo major surgery that will have an impact on their subsequent quality of life. Preparing for this surgery is a lengthy process, involving various forms of support: psychological, nutritional, physical activity, and so on. Exploring patients' experiences in depth, based on their account of their care experience, can enable carers to better understand and apprehend this type of journey from a perspective closer to that of the patient.

DETAILED DESCRIPTION:
Given the growing importance of placing the patient at the heart of care evaluation, the use of patient questionnaires such as Patient Reported Experience Measures (PREMS) or Patient-Reported Outcome Measures (PROMS) has become widespread in recent years. PROMS assess the outcomes of care, whereas PREMS assess the patient's experience of care. However, these tools only imperfectly reflect the patient's experience and only answer specific questions: satisfaction, pain management, waiting times, etc. Other initiatives, such as the patient tracer (https://www.has-sante.fr/jcms/c_2807803/fr/patient-traceur), involve interviewing patients and, where appropriate, their relatives about their care by asking them specific questions about their care, such as the information they have received, the therapeutic workshops they have attended, etc. However, all these attempts to put the patient at the centre of the evaluation of the quality of care are still based on quality questions or indicators defined a priori by healthcare professionals and the health authorities.

Patients undergoing bariatric surgery will undergo major surgery that will have an impact on their subsequent quality of life. Preparing for this surgery is a lengthy process, involving various forms of support: psychological, nutritional, physical activity, and so on. Exploring patients' experiences in depth, based on their account of their care experience, can enable carers to better understand and apprehend this type of journey from a perspective closer to that of the patient.

The narrative inquiry method enables patients' unique experiences to be collected and co-constructed with the help of interviewers. In addition, this qualitative approach focuses not only on the experience of individuals, but also on the social and cultural aspects in which they are embedded, enabling a more global and less reductive approach to the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient enrolled in a bariatric surgical pathway scheduled.
* First bariatric surgery

Exclusion Criteria:

* Refusal to participate
* Non proficiency in spoken French
* Previous bariatric surgery
* Protected persons (patients under guardianship, pregnant or breastfeeding women, persons deprived of liberty, persons unable to express their non-objection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
patient experience of the care pathway | 6 months
  Explain the bariatric surgery care pathway, based on the patient experience

SECONDARY OUTCOMES:
Questionnaire | 3 months
  Construction of a questionnaire based on the common meta-narrative
Number of experiences collected | 3 months
  Number of complete patient experiences collected
Repeat surgeries | 3 months
  Number of repeat surgeries for up to 3 months after surgery
Repeat hospitalizations | 3 months
  Number of repeat hospitalizations for up to 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vignot M, Jung C, Bathaei S, Lazzati A, Gateau V, Angeli F, Delorenzo C. Patient experience in bariatric surgery: protocol of a French narrative inquiry and qualitative analysis. BMJ Open. 2024 Aug 12;14(8):e082528. doi: 10.1136/bmjopen-2023-082528. PMID 39134437